CLINICAL TRIAL: NCT00087399
Title: A Phase III Randomized, Trial of Gabapentin Alone or in Conjunction With an Antidepressant in the Management of Hot Flashes in Women Who Have Inadequate Control With an Antidepressant Alone
Brief Title: Gabapentin With or Without Antidepressants in Treating Hot Flashes in Women Who Have Had Breast Cancer or Have Concerns About Taking Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCCTG-N03C5; NCI-2012-02616 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000374993 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Hot Flashes
Keywords: breast cancer; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Gabapentin; Antidepressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gabapentin + antidepressant (Experimental): Patients continue to receive the same antidepressant (as before study entry) on weeks 1-5. During weeks 2-5, patients also receive oral gabapentin once daily on days 8-10, twice daily on days 11-13, and then three times daily on days 14-35 in the absence of unacceptable toxicity.
  Patients complete a hot flash diary at baseline and then daily during study treatment.
  Interventions: Drug: gabapentin; Drug: antidepressant
- gabapentin (Experimental): Patients receive gabapentin once daily on days 8-10, twice daily on days 11-13, and then three times daily on days 14-35 in the absence of unacceptable toxicity. Patients are tapered off their antidepressant over 7-10 days and remain on gabapentin alone.
  Patients complete a hot flash diary at baseline and then daily during study treatment.
  Interventions: Drug: gabapentin

INTERVENTIONS:
Drug: gabapentin
Drug: antidepressant
  Arms: gabapentin + antidepressant

SUMMARY:
RATIONALE: Gabapentin may be effective in relieving hot flashes in women who have had breast cancer or who have concerns about taking hormone therapy to treat hot flashes. It is not yet known whether gabapentin is more effective with or without antidepressants in treating hot flashes.

PURPOSE: This randomized phase III trial is studying gabapentin and antidepressants to see how well they work compared to antidepressants alone in treating hot flashes in women who have had breast cancer or who have concerns about taking hormones to treat hot flashes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of gabapentin with vs without an antidepressant, as measured by the frequency and intensity of hot flashes, in patients with a history of breast cancer or a concern about taking hormonal therapy due to a fear of developing breast cancer.
* Compare adverse events in patients treated with these regimens.
* Correlate a reduction in hot flash scores with improvement in quality of life and related outcomes in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to duration of hot flash symptoms (< 9 months vs ≥ 9 months), average frequency of hot flashes per day (2-3 vs 4-9 vs ≥ 10), and antidepressant currently being used (venlafaxine vs paroxetine vs other). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients continue to receive the same antidepressant (as before study entry) on weeks 1-5. During weeks 2-5, patients also receive oral gabapentin once daily on days 8-10, twice daily on days 11-13, and then three times daily on days 14-35 in the absence of unacceptable toxicity.
* Arm II: Patients receive gabapentin as in arm I. Patients are tapered off their antidepressant over 7-10 days and remain on gabapentin alone (per arm I schedule).

Patients in both arms complete a hot flash diary at baseline and then daily during study treatment.

Quality of life is assessed at baseline and then weekly during study treatment.

PROJECTED ACCRUAL: A total of 110 patients (55 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of breast cancer OR a concern about taking hormonal therapy due to a fear of developing breast cancer
* Experiencing bothersome hot flashes, defined as patient-reported occurrence ≥ 14 times per week AND sufficiently severe to prompt desire for additional therapeutic intervention despite current use of an antidepressant

  * Currently (≥ 2 weeks) being treated with a stable dose of an antidepressant

    * No monoamine oxidase inhibitors or tricyclics
* No current evidence of malignant disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Performance status

* ECOG 0-1

Life expectancy

* At least 6 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Chemotherapy

* More than 4 weeks since prior antineoplastic chemotherapy
* No concurrent antineoplastic chemotherapy

Endocrine therapy

* More than 4 weeks since prior androgens, estrogens, or progestational agents
* More than 2 weeks since prior dehydroepiandrosterone (DHEA) for treatment of hot flashes
* No concurrent androgens, estrogens, or progestational agents, including oral contraceptives
* No concurrent DHEA for treatment of hot flashes
* Concurrent tamoxifen, raloxifene, or aromatase inhibitor therapy allowed if on a stable dose for at least 4 weeks prior to study entry and during study treatment

Other

* No prior gabapentin
* More than 2 weeks since other prior treatment for hot flashes (e.g., clonidine or Bellergal-S®)
* Concurrent vitamin E or soy supplements allowed if on a stable dose for at least 1 month prior to study entry and during study treatment
* No other concurrent treatment for hot flashes (e.g., clonidine or Bellergal-S®)
* No other concurrent antidepressants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Hot flash reduction by diary record at 4 weeks | at 4 weeks

SECONDARY OUTCOMES:
Toxicity by questionnaires at 4 weeks | at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (162):
- United States (162):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Alegent Health Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Cancer Center at Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Mercy and Unity Hospitals, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Saint Cloud, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - Cancer Care Center at Regions Hospital, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Hospital, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Cancer Center at Creighton University Medical Center, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Health System, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - Guthrie Medical Center - Sayre, Sayre, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Loprinzi CL, Kugler JW, Barton DL, Dueck AC, Tschetter LK, Nelimark RA, Balcueva EP, Burger KN, Novotny PJ, Carlson MD, Duane SF, Corso SW, Johnson DB, Jaslowski AJ. Phase III trial of gabapentin alone or in conjunction with an antidepressant in the management of hot flashes in women who have inadequate control with an antidepressant alone: NCCTG N03C5. J Clin Oncol. 2007 Jan 20;25(3):308-12. doi: 10.1200/JCO.2006.07.5390. Epub 2006 Dec 4. PMID 17146104
- [Result] Loprinzi CL, Kugler JW, Barton DL, et al.: Phase III randomized trial to evaluate the use of gabapentin alone vs with continuing an antidepressant in women failing an antidepressant for the treatment of hot flashes: North Central Cancer Treatment Group study N03C5. [Abstract] J Clin Oncol 24 (Suppl 18): A-526, 9s, 2006.